CLINICAL TRIAL: NCT02847429
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial of Crenolanib in Subjects With Advanced or Metastatic Gastrointestinal Stromal Tumors With a D842V Mutation in the PDGFRA Gene
Brief Title: Randomized Trial of Crenolanib in Subjects With D842V Mutated GIST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arog Pharmaceuticals, Inc. (Industry)
Collaborators: Centre Leon Berard (Other); Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARO-012; 2015-000287-34 (EudraCT Number)
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: GIST With D842V Mutated PDGFRA Gene
MeSH Terms: interventions — crenolanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crenolanib Arm (Experimental): Investigational product (crenolanib)
  Interventions: Drug: Crenolanib
- Placebo Arm (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Crenolanib
  Other Names: Crenolanib Besylate
  Arms: Crenolanib Arm
Drug: Placebo
  Arms: Placebo Arm

SUMMARY:
This is a multicenter, randomized, double-blinded, placebo-controlled, trial of oral crenolanib versus oral placebo in combination with best supportive care in subjects with advanced or metastatic GIST with a D842V mutation in the PDGFRA gene. Approximately 120 subjects will be randomized in a 2:1 ratio to receive either crenolanib 100 mg or matching placebo orally (PO) 3 times daily (TID) in combination with best supportive care.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically-confirmed advanced or metastatic GIST with a D842V mutation in the PDGFRA gene as determined by central laboratory testing
2. Measurable disease as per modified RECIST 1.1

   • A lesion in an area that was previously treated with local therapy (e.g. radiation, surgery, or cryotherapy) can be considered measurable disease as long as there is objective evidence of progression of the lesion prior to randomization
3. Subjects (male or female) ≥ 18 years of age
4. Female subjects with reproductive potential must have negative serum or urine pregnancy test
5. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2

Exclusion Criteria:

1. Severe liver disease (e.g. cirrhosis, non-alcoholic steatohepatitis, sclerosing cholangitis)
2. Known, active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
3. Female subject who is pregnant or breastfeeding, or planning to become pregnant within 30 days after ending treatment
4. Systemic anti-cancer treatment (e.g. chemotherapy, tyrosine kinase inhibitors, immunotherapy, or investigational agents) or investigational device within 3 weeks or 5 half-lives (if the drug's half-life in subject is known) prior to randomization, whichever is shorter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-08; Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) will be measured from the date of randomization to the date of the first objective radiological disease progression according to centralized committee assessment using modified RECIST version 1.1 or death. | 3 years

SECONDARY OUTCOMES:
Overall survival (OS) will be measured from the date of randomization to the date of death from any cause. OS will be estimated using the Kaplan-Meier method. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Blay, MD, Principal Investigator — Centre Leon Berard; Margaret von Mehren, MD, Principal Investigator — Fox Chase Cancer Center
Locations (23):
- United States (6):
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Miami, Miami, Florida
  - Duke Cancer Institute, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- France (4):
  - Institut Bergonie, Bordeaux
  - Centre Leon Berard, Lyon
  - La Timone University Hospital, Marseille
  - Centre Hospitalier Universitaire (CHU) de Reims, Reims
- Germany (3):
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Mannheim University Medical Centre, University of Heidelberg, Mannheim
  - Universitätsklinikum München, Munich
- Italy (4):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Istituto Nazionale Tumori, Milan
  - Institut Regina Elena / IFO, Rome
  - Candiolo Cancer Institute - FPO, IRCCS, Turin
- University Hospital The Norwegian Radium Hospital, Oslo, Norway
- M Sklodowska-Curie Memorial Cancer Centre and Institute of Oncology, Warsaw, Poland
- Spain (4):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Virgen del Rocio, Seville
  - Fundación Instituto Valenciano de Oncología, Valencia